CLINICAL TRIAL: NCT06069986
Title: On-pump Versus Off-pump Coronary Artery Bypass Grafting , Short Term Outcomes , Sohag Experience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ziad Essam Ahmed, assistant lecturer cardithoracic surgery sohag university, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-09-1MD
Record Dates: First submitted 2023-09-13; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- on pump CABG (Active Comparator): using cardiopulmonary bypass
  Interventions: Procedure: coronary artery bypass graft CABG
- off pump CABG (Active Comparator): without cardiopulmonary bypass
  Interventions: Procedure: coronary artery bypass graft CABG

INTERVENTIONS:
Procedure: coronary artery bypass graft CABG — comparison between onpump and off pump CABG

SUMMARY:
Coronary artery disease (CAD) and its sequlae, such as myocardial infarction, arrhythmia and heart failure, are among the leading causes of death around the world . the durable role of coronary artery bypass grafting (CABG) in the treatment of CAD has long been shown.

Coronary artery bypass grafting (CABG) is a commonly performed surgical procedure for patients with coronary artery disease (CAD), CABG can be performed using either the on-pump or off-pump technique, each with its own advantages and limitations.

On-pump CABG involves the use of CPB which as agold standard for surgical coronary revascularization has led toexcellent results in mortality and complications. On-pump CABG allows the surgeon to temporarily stop the heart and provide perfusion and oxygenation to the body. This technique provides a bloodless and motionless operative field, allowing for precise graft anastomosis. However, the use of CPB is associated with deleterious effects as systemic inflammatory response, hemodilution, and organ dysfunction as dysrhythmia and neurocognitive problems. These factors may adversely affect patients lives specially those with impaired EF, who already have compromised cardiovascular function.

Another technique for CABG is on-pump beating heart CABG (ONBH-CABG) surgery that is relatively novel hybrid approach to coronary artery grafting which aims to stabilize hemodynamic parameters during the operative period. This has specific benefits such as reduced preload alongside the afterload which decreases the oxygen demand of the myocardial tissue

ELIGIBILITY:
Inclusion Criteria:

* fair and impaired EF

Exclusion Criteria:

* malignancy
* COPD
* renal failure on dialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
comparison to declare the rate of morbidity and mortality using both techniques on pump and off pump in CABG and which is better in short term outcomes | 1 year
  which is better in morbidity and mortality, on pump or off pump CABG specially in patients with low ejection fraction (less than 40%)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lamy A, Devereaux PJ, Prabhakaran D, Taggart DP, Hu S, Paolasso E, Straka Z, Piegas LS, Akar AR, Jain AR, Noiseux N, Padmanabhan C, Bahamondes JC, Novick RJ, Vaijyanath P, Reddy S, Tao L, Olavegogeascoechea PA, Airan B, Sulling TA, Whitlock RP, Ou Y, Ng J, Chrolavicius S, Yusuf S; CORONARY Investigators. Off-pump or on-pump coronary-artery bypass grafting at 30 days. N Engl J Med. 2012 Apr 19;366(16):1489-97. doi: 10.1056/NEJMoa1200388. Epub 2012 Mar 26. PMID 22449296
- [Background] Ascione R, Narayan P, Rogers CA, Lim KH, Capoun R, Angelini GD. Early and midterm clinical outcome in patients with severe left ventricular dysfunction undergoing coronary artery surgery. Ann Thorac Surg. 2003 Sep;76(3):793-9. doi: 10.1016/s0003-4975(03)00664-7. PMID 12963202
- [Background] Ueki C, Miyata H, Motomura N, Sakaguchi G, Akimoto T, Takamoto S. Off-pump versus on-pump coronary artery bypass grafting in patients with left ventricular dysfunction. J Thorac Cardiovasc Surg. 2016 Apr;151(4):1092-8. doi: 10.1016/j.jtcvs.2015.11.023. Epub 2015 Nov 22. PMID 26725715
- [Background] Shroyer AL, Hattler B, Wagner TH, Collins JF, Baltz JH, Quin JA, Almassi GH, Kozora E, Bakaeen F, Cleveland JC Jr, Bishawi M, Grover FL; Veterans Affairs ROOBY-FS Group. Five-Year Outcomes after On-Pump and Off-Pump Coronary-Artery Bypass. N Engl J Med. 2017 Aug 17;377(7):623-632. doi: 10.1056/NEJMoa1614341. PMID 28813218